CLINICAL TRIAL: NCT03864315
Title: To Study the Efficacy of Therapeutic Pulsed Ultrasound in the Treatment of Vitiligo: a Randomized, Intra-individual, Left-right Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201403043DINC
Record Dates: First submitted 2019-02-25; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Vitiligo
Keywords: Vitiligo; Harmonic Generation Microscopy; In Vivo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitiligo (Experimental): 30 Patients with Vitiligo
  Interventions: Device: HGM

INTERVENTIONS:
Device: HGM — To Study the Efficacy of Therapeutic Pulsed Ultrasound in the Treatment of Vitiligo: a Randomized, Intra-individual, Left-right Comparison Study

SUMMARY:
In this study, the investigators demonstrated that in vivo THG microscopy can differentiate vitiligo lesions and normal skin based the optical nature of melanin. This THG-based procedure provides a valuable tool for noninvasive determination of third-order nonlinear susceptibility of melanin within the skin. It can also provide real-time histopathology information for treatment follow-up, without performing invasive skin biopsy.

DETAILED DESCRIPTION:
The investigators initiate this open, randomized, left-right comparative study to evaluate the efficacy of pulsed ultrasound in the treatment of vitiligo on the face or trunk. Face is included in this study because vitiliginous lesions on the face has a better treatment response and causes more psychological distress on the patients than vitiligo affecting other body areas. Thirty adult subjects with vitiligo affecting the face or trunk symmetrically will be recruited. After randomization, subjects will be administrated their ulrasound treatment twice a week for 24 weeks. Their original topical treatment and/or phototherapy will be continued. During follow-up visits, digital photographs will be taken for evaluating the extent of residual depigmentation. In vivo harmonic microscopy and three skin biopsy specimens will be performed at the indicated time points on the depigmented, repigmented areas and surrounding normal skin.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75 years old
2. With skin type Ⅲ or Ⅳ
3. With Vitiligo
4. Can read the informed consent form
5. Can continue the original treatments

Exclusion Criteria:

1. With segmental vitiligo.
2. Have joined other clinical trials

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2014-10-23 (Actual); Study Completion 2015-12-09 (Actual)

PRIMARY OUTCOMES:
30 participants with Vitiligo as assessed by Harmonic Generation Microscopy. | 1-2 hours per case
  The HGM system will be combined to provide the noninvasive microscopic images in Vitiligo sites during each follow-up for pathological diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan